CLINICAL TRIAL: NCT00290121
Title: Cerebral Mechanism Involved in Appetite Increase in Schizophrenia Patients Treated With Atypical Antipsychotics (IIT)
Brief Title: Appetite Increase in Schizophrenia Patients Treated With Atypical Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other); Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2005-0503
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2005-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Atypical antipsychotics; Weight gain; Appetite; fMRI
MeSH Terms: conditions — Schizophrenia; Weight Gain | interventions — Olanzapine

ARMS (1):
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
The purpose of this study is to understand, with the use of functional magnetic resonance imaging, the neural correlates involved in appetite control and the mechanism of weight gain in patients with schizophrenia treated with atypical antipsychotics. We hypothesize that a difference in cerebral activations between weight gaining and non-weight gaining patients will be detected after four months of treatment with olanzapine.

DETAILED DESCRIPTION:
Atypical antipsychotics (AAP) have revolutionize treatment of schizophrenia. They are considered to be more effective in reducing positive and negative symptoms and in improving cognitive deficits. They cause less extrapyramidal symptoms and tardive dyskinesia than typical antipsychotics. They still have a lot of important side effects like sedation, metabolic syndrome and weight gain. These effects could lead to obesity, type II diabetes and cardiovascular diseases, particularly for schizophrenia patients because they are already at an increased risk for these complications. Moreover, an increase in weight gain has been demonstrate to exacerbate negative symptoms and can lead to non compliance with a consequent risk of relapse. It also can create an additional social disadvantage for schizophrenia patients and decrease their quality of life. The weight gain will result, in part from an increased food intake (and probably an increased appetite) and from a decreased energy expenditure.

The purpose of this study is to understand the cerebral mechanisms of appetite in patients with schizophrenia treated with atypical antipsychotics to prevent or treat their weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia (DMS-IV)
* 18 to 60 years old
* Right handed
* Begin a treatment with olanzapine and had not received it for at leat 6 months
* Other medication accepted (except antipsychotic)

Exclusion Criteria:

* concomitant axis-I or axis-II disorders
* unstable medical condition
* Concomitant antipsychotic medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
fMRI (functional magnetic resonance imaging with appetizing films) | 16 weeks after beginning of Olanzapine treatment
Weight | 16 weeks after beginning of Olanzapine treatment

SECONDARY OUTCOMES:
Fasting glucose | 16 weeks after beginning of Olanzapine treatment
Insulin | 16 weeks after beginning of Olanzapine treatment
Leptin | 16 weeks after beginning of Olanzapine treatment
Ghrelin | 16 weeks after beginning of Olanzapine treatment
Endogenous cannabinoids | 16 weeks after beginning of Olanzapine treatment
Lipid profile | 16 weeks after beginning of Olanzapine treatment
PANSS (Positive and negative syndrome scale) | 16 weeks after beginning of Olanzapine treatment
CDSS (Calgary Depression scale for schizophrenia) | 16 weeks after beginning of Olanzapine treatment
Three factors eating questionnaire | 16 weeks after beginning of Olanzapine treatment
Fagerstrom test for nicotine dependence | 16 weeks after beginning of Olanzapine treatment
Adult ADHD (attention deficit hyperactivity disorder) self report scale | 16 weeks after beginning of Olanzapine treatment
Age | 16 weeks after beginning of Olanzapine treatment
Sexe | 16 weeks after beginning of Olanzapine treatment
Weight | 16 weeks after beginning of Olanzapine treatment
Abdominal circumference | 16 weeks after beginning of Olanzapine treatment
Number and times of hospitalization | 16 weeks after beginning of Olanzapine treatment
Blood pressure | 16 weeks after beginning of Olanzapine treatment
Prolactin | 16 weeks after beginning of Olanzapine treatment
Onset of disease | 16 weeks after beginning of Olanzapine treatment
Level of education | 16 weeks after beginning of Olanzapine treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Stip, MD, M.Sc., Principal Investigator — Centre de recherche Fernand-Seguin, Université de Montréal
Locations (1):
- Centre de recherche Fernand-Seguin, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Orban P, Desseilles M, Mendrek A, Bourque J, Bellec P, Stip E. Altered brain connectivity in patients with schizophrenia is consistent across cognitive contexts. J Psychiatry Neurosci. 2017 Jan;42(1):17-26. doi: 10.1503/jpn.150247. PMID 27091719
- [Derived] Stip E, Lungu OV. Salience network and olanzapine in schizophrenia: implications for treatment in anorexia nervosa. Can J Psychiatry. 2015 Mar;60(3 Suppl 2):S35-9. PMID 25886678
- [Derived] Stip E, Lungu OV, Anselmo K, Letourneau G, Mendrek A, Stip B, Lipp O, Lalonde P, Bentaleb LA. Neural changes associated with appetite information processing in schizophrenic patients after 16 weeks of olanzapine treatment. Transl Psychiatry. 2012 Jun 19;2(6):e128. doi: 10.1038/tp.2012.53. PMID 22714121